CLINICAL TRIAL: NCT04664504
Title: A Prospective Phase II Study of Individualized Neoadjuvant Chemoradiotherapy for Rectal Cancer Based on Recurrence Risk
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jing Jin, M.D. (Unknown)
Responsible Party: Sponsor-Investigator, Jing Jin, M.D., Clinical Professor, Radiotherapy Department, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3332019055
Record Dates: First submitted 2020-12-06; First posted 2020-12-11 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Rectal Cancer
Keywords: Rectal Cancer; Neoadjuvant Chemoradiotherapy; Recurrence Risk
MeSH Terms: conditions — Rectal Neoplasms | interventions — Consolidation Chemotherapy; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group CRT (Active Comparator): concurrent chemoradiotherapy → TME → adjuvant chemotherapy (control group)
  Interventions: Combination Product: Concurrent Chemoradiotherapy Radiotherapy; Drug: Adjuvant chemotherapy; Procedure: TME
- Group SCRT (Experimental): Short-course radiotherapy→ consolidation chemotherapy → TME (experimental group)
  Interventions: Radiation: Short-course Radiotherapy; Drug: Consolidation chemotherapy; Procedure: TME
- Group es-SCRT (Experimental): Local dose increase of Short-course radiotherapy→ consolidation chemotherapy → TME (experimental group)
  Interventions: Radiation: Local dose increase of Short-course Radiotherapy; Drug: Consolidation chemotherapy; Procedure: TME

INTERVENTIONS:
Combination Product: Concurrent Chemoradiotherapy Radiotherapy — 50Gy in 25 fractions to the primary tumor and to mesorectal, presacral,and internal iliac lymph nodes. Concurrent chemotherapy: Capecitabine 1650 mg/m2/d.
  Other Names: CRT
  Arms: Group CRT
Radiation: Short-course Radiotherapy — 25Gy in 5 fractions to the primary tumor and to mesorectal, presacral,and internal iliac lymph nodes.
  Other Names: SCRT
  Arms: Group SCRT
Radiation: Local dose increase of Short-course Radiotherapy — 25Gy in 5 fractions to the of primary tumor and to mesorectal, presacral,and internal iliac lymph nodes. And 4Gy in 1 fractions to the PGTV of primary tumor and to mesorectal, presacral,and internal iliac lymph nodes.
  Other Names: es-SCRT
  Arms: Group es-SCRT
Drug: Consolidation chemotherapy — Intravenous infusion of oxaliplatin (130 mg/m2 over 2 h) on day 1 and oral administration of capecitabine (1000 mg/m2 twice daily) from day 1 to day 14, is repeated every 3 weeks for 4 cycles. 4 courses*3 weeks per course.
  Other Names: XEOLX*4 courses
  Arms: Group SCRT; Group es-SCRT
Drug: Adjuvant chemotherapy — 2 h) on day 1 and oral administration of capecitabine (1000 mg/m2 twice daily) from day 1 to day 14, is repeated every 3 weeks for 6 cycles. 6 courses*3 weeks per course
  Other Names: XEOLX*6 courses
  Arms: Group CRT
Procedure: TME — Total mesorectal excision

SUMMARY:
A Prospective Phase II Study of Individualized Neoadjuvant Chemoradiotherapy for Rectal Cancer Based on Recurrence Risk

DETAILED DESCRIPTION:
For patients with locally advanced rectal cancer, radiotherapy and chemotherapy combined with surgery can improve the curative effect. Rectal magnetic resonance imaging (MRI) can be used to stratify the risk of locally advanced rectal cancer before treatment. In this study, we planned to use rectal MRI parameters and the possibility of patients with anal preservation to group, and to observe the R0 resection rate and disease-free survival rate of patients with stage II / III rectal cancer after individualized preoperative radiotherapy and chemotherapy combined with radical surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Rectal adenocarcinoma confirmed by histopathology
2. MRI staging was stage II / III (cT3-T4N0 or cT2-4N+)
3. The age is 18-75 years old, no gender limit

3) The distance between the lower limit of the lesion and the anal margin was less than or equal to 10 cm 4) Karnofsky score ≥ 80 or ECOG score 0-1

Exclusion Criteria:

1. History of other malignant tumors;
2. They were allergic to 5-FU, platinum, etc;
3. The patient is in thrombolytic and anticoagulant therapy, and has bleeding quality or coagulation dysfunction; or in the past year, aneurysm, stroke, transient ischemic attack, arteriovenous malformation occurred;
4. After the previous renal history, proteinuria or clinical renal function were found to be abnormal;
5. History of gastrointestinal fistula, perforation or severe ulcer;
6. At present, there are active infection; clinical obvious heart disease; New York Heart Association (NYHA) ≥ grade II congestive heart failure; unstable symptomatic arrhythmia or peripheral vascular disease ≥ grade II; myocardial infarction and cerebrovascular accident occurred within 6 months before enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | 1 year
  R0 resection rate is R0 resection probability of radical surgery in patients with locally advanced rectal cancer after individualized chemoradiotherapy

SECONDARY OUTCOMES:
3y OS | 3 years
  3-year overall survival
3yDMFS | 3 years
  3-year distant metastatic free survival
3yLRRFS | 3 years
  3-year locoregional recurrence-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Tang, M.D., Study Director — Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Department of Radiation Oncology, Cancer Institute and Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Beijing, China